CLINICAL TRIAL: NCT01233986
Title: Prospective, Matched Case Control, Multicenter, Observational Study for the Association of Serum Apolipoprotein B-48 Level and Large arterY Atherosclerotic iSchemic Stroke(ABYSS)
Brief Title: Association of Apolipoprotein B-48 Level and Large arterY Atherosclerotic iSchemic Stroke(ABYSS)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hallym University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: ABYSS
Record Dates: First submitted 2010-10-21; First posted 2010-11-04 (Estimated); Last update posted 2011-10-05 (Estimated); Status verified 2010-11

CONDITIONS: Acute Ischemic Stroke
Keywords: Acute Ischemic Stroke; Atherosclerosis; Apolipoprotein B48
MeSH Terms: conditions — Ischemic Stroke; Atherosclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum level of apolipoprotein B-48
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Case group - Large artery atherosclerosis
- Control group-Small vessel occlusion

SUMMARY:
The purpose of this study is to evaluate whether the serum apoB48 level is associated with atherosclerotic ischemic stroke.

ELIGIBILITY:
Inclusion Criteria:

Large artery atherosclerotic ischemic stroke group(LAA group)

* Age over 20 years
* Patients with symptomatic stenosis in the eligible vessels(the middle cerebral artery, anterior cerebral artery, or internal carotid artery) as assessed by MRA or CTA corresponding to the acute ischemic stroke
* Patients without the occlusion of corresponding artery by MRA or CTA
* The fasting and postprandial serum Apo B-48 level can be assessed within 72 hours after the symptom onset of ischemic stroke

Small vessel occlusive ischemic stroke group (SVO group)

* Age over 20 years
* Patients with acute ischemic stroke of basal ganglia, internal capsule, or corona radiata
* Patients without both symptomatic and asymptomatic arterial occlusion or stenosis by MRA or CTA
* Patients without a history of systemic atherosclerosis(for example, acute myocardial infarction, angina, peripheral arterial disease, aortic aneurysm)
* The fasting and postprandial serum Apo B-48 level can be assessed within 72 hours after the symptom onset of ischemic stroke

Exclusion Criteria: both LAA group and SVO group

* Patients with cardioembolic ischemic stroke
* Patients treated with lipid lowering agents or steroid within the previous 30 dsys
* Patients with severe liver disease (AST >100 or ALT >100) at the time of randomization
* Patients with endocrine disease except diabetes mellitus at the time of randomization (for example, thyroid disease, adrenal disease)
* Patients with severe renal disease (serum creatinine >2.0mg/dl)at the time of randomization
* chronic alcoholics or drug user
* Patients with infection at the time of randomization
* Patients, in the opinion of the investigator, unlikely to comply with the clinical study or unsuitable for the any other disease or reason
* Informed consent has not been obtained

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Tertiary Hospital
Sampling Method: Probability Sample
Enrollment: 112 (Estimated)
Dates: Start 2010-05; Primary Completion 2011-03 (Actual); Study Completion 2011-10 (Estimated)

PRIMARY OUTCOMES:
The serum level of fasting apolipoprotein B-48 | 72 hours within stroke onset
The serum level of postprandial apolipoprotein B-48 | within 72 hours after stroke onset

SECONDARY OUTCOMES:
The serum level of the postprandial triglyceride | 72 hours within stroke onset
The serum level of fasting total cholesterol | within 72 hours after stroke onset
The serum level of fasting LDL cholesterol | within 72 hours after stroke onset
the level of fasting HDL cholesterol | within 72 hours after stroke onset
the level of fasting triglyceride | within 72 hours after stroke onset

CONTACTS AND LOCATIONS:
Overall Officials: Byung-Chul Lee, MD,PhD, Principal Investigator — Hallym University Medical Center
Locations (1):
- Hallym University Sacred Heart Hospital, Anyang, Anyang, South Korea